CLINICAL TRIAL: NCT03536533
Title: Effects of a Virtual Reality-based Dual-task Exercise on Vestibular Function in Patients With Chronic Peripheral Unilateral Vestibular Hypofunction
Brief Title: Virtual Reality-based Dual-task Exercise in Vestibular Hypofunction Patients
Acronym: VR-VH-ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2018-00337
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Vestibular Diseases
MeSH Terms: conditions — Vestibular Diseases | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergame (Experimental): The Senso is a training system (dividat, Schindellegi, Switzerland) for improving physical and cognitive function was used as exergame. With foot pushes participants triggered on a pressure-sensitive plate. The Senso game was projected with a beamer at white wall. To promote head movement during training the direction of the beamer was vertical tilted (± 15°) and horizontal turned (90°) with a remote controlled power panner.
  Interventions: Other: Exergame

INTERVENTIONS:
Other: Exergame — Each of the 8 exercise sessions will last at least 42 minutes, with an actual training duration of 21 minutes. The participants will be accustomed gradually to the game. On one hand this will be achieved by increasing the difficulty in subsequent levels within the exergame.
  Other Names: SENSO Dividat

SUMMARY:
The aim is to assess the effects of virtual reality-based intervention on vestibular functions in in patients with chronic peripheral unilateral vestibular hypofunction.

DETAILED DESCRIPTION:
In a close interplay of sensory and motor functions, the brain constantly evaluates intrinsic and extrinsic movements, creating an inner - always subjective - representation of the stability. If there is an acute or chronic imbalance ("mismatch"), a multisensory misperception can occur. This is perceived subjectively as dizziness. Dizziness is the third most common neurological cause of an emergency with 11-13% after headache and stroke.

The central vestibular system is often involved in dizziness. The organ is part of the inner ear and is located in the petrous bone. It consist of macula organs, which are responsible for the detection of linear accelerations, and semicircular canals, which perceive the head velocity. Furthermore, the central vestibular system provides ocular muscles and the spinal cord with output, in order to control three reflexes. The vestibulo-ocular reflex (VOR) is responsible for a clear vision while the head is rotating, whereas the vestibulo-collic reflex (VCR) innervates the neck musculature in order to fix the head. The purpose of the vestibulo-spinal reflex (VSR) is the stabilization of the body by compensatory movements. In terms of restoring vestibular functioning, compensation can be classified into adaptation, substitution and habituation. Adaptation enhances the VOR, which is equivalent to restoration. Substitution is distinguished in literature between sensory and behavioral, in which the sensorial substitution transfers the importance given to proprioceptive and visual inputs and the behavioral substitution refers to avoidance strategies e.g. immobilization, increased blink reflex and prevention of head rotations. Habituation on the other hand, accustoms the affected person to a conflicting situation, in order that the response of the VOR is avoided.

So far, it is known that previous conventional vestibular rehabilitation is effective for age-related vestibular loss. By improving vestibular function, the vestibular rehabilitation therapy aims to improve balance and neuromuscular coordination, minimize falls and decrease the feeling of dizziness.

However, new advances in technology have been made which generate additional methods for an effective therapy; exercise and videogaming, in short, exergaming. Successful use of virtual reality in rehabilitation of vestibular patients has previously been implemented. Further, recent evidence has examined the effects of exergaming in healthy dwellers on vestibular function. There was a significant reduction found in the dynamic visual acuity (DVA) after an eight-session exergame training (in total 160 minutes).

To date, the effects on vestibulo-ocular reflex of exergames in patients with chronic peripheral vestibular hypofunction have not been systematically explored. Moreover, very little is known about the effects of exergaming includes exercises requiring head turns on vestibular function in this patients. Furthermore, exergaming could become a new tool to improve DVA and dizziness and increase the training intensity without requiring many therapists, which in turn reduces health costs. In addition, patients with dizziness are severely affected by their disease. They will welcome new, efficient and motivating forms of therapy.Finally, the main aim is to assess the effects of virtual reality-based intervention with dividat "senso" on vestibular functions in patients with chronic peripheral unilateral vestibular hypofunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic peripheral unilateral vestibular hypofunction
* Signed informed consent after being informed

Exclusion Criteria:

* Patients with Benign paroxysmal positional vertigo and/or Menière's disease
* Walking disability (independent walking <10 meters)
* Acute pain and limited range of motion in cervical spine
* Gait disorders putatively attributed to other than primarily vestibular causes
* Weakness due to neurological problems
* Uncontrolled cardiovascular disease
* Medication reducing postural balance
* Uncorrected heavy visual impairment
* Acute pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Visual Acuity (DVA) | 15 minutes
  The DVA is the measurement of visual acuity during head movement relative to baseline static visual acuity

SECONDARY OUTCOMES:
Video Head Impulse Test (vHIT) | 15 minutes
  The vHIT will be used to test the vestibulo-ocular reflex.
Suppression Head Impulse Paradigm (SHIMP) | 15 minutes
  In contrary to vHIT, which indicate a compensatory saccade and thus a vestibular loss, the suppression head impulse paradigm (SHIMP) measures the vestibular function
Subjective Visual Vertical test (SVV) | 15 minutes
  SVV assesses the ability to perceive verticality which depends on input from visual, somatosensory and vestibular system
Functional Gait Assessment (FGA) | 15 minutes
  The FGA is used to measure disturbances in balance and gait
Extended Timed Get-Up-And-Go (ETGUG) | 15 minutes
  The time measured during each task and the overall time mirrors the functional mobility of the participant
Simulator Sickness Questionnaire (SQQ) | 5 minutes
  The SSQ questionnaire assesses, cyber or virtual reality sickness
Misery Score (MISC 1-6) | 1 minutes
  The Misery score is a scale to gather the nausea symptom
Dizziness handicap inventory (DHI) | 10 minutes
  The DHI is questionnaire to evaluate the self-perceived handicapping effects caused by dizziness
Game Scores | 1 minutes
  Game intervention administration and dosage (frequency, intensity, time and type of the video game

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research
Locations (1):
- University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No